CLINICAL TRIAL: NCT03816670
Title: Prospective Randomized Trial Comparing Corifollitropin-alfa Late Start (Day 4) vs. Corifollitropin-alfa Standard Start (Day 2) in Expected Poor, Normal and High-responders Undergoing IVF/ICSI
Brief Title: Prospective Randomized Trial Comparing Corifollitropin-alfa Late Start vs. Corifollitropin-alfa Standard Start in Expected Poor, Normal and High-responders Undergoing IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Alberto Revelli, Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIS#53736
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Fertility Disorders
MeSH Terms: interventions — follicle stimulating hormone, human, with HCG C-terminal peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- poor responders day 2 (Experimental): "poor responders" women stimulated with CF from day 2 of menstrual cycle
  Interventions: Drug: Corifollitropin Alfa
- poor responders day 4 (Experimental): "poor responders" women stimulated with CF from day 4 of menstrual cycle
  Interventions: Drug: Corifollitropin Alfa
- normal responders day 2 (Experimental): "normal responders" women stimulated with CF from day 2
  Interventions: Drug: Corifollitropin Alfa
- normal responders day 4 (Experimental): "normal responders" women stimulated with CF from day 4
  Interventions: Drug: Corifollitropin Alfa
- high responders day 2 (Experimental): "high responders" women stimulated with CF from day 2
  Interventions: Drug: Corifollitropin Alfa
- high responders day 4 (Experimental): "high responders" women stimulated with CF from day 4
  Interventions: Drug: Corifollitropin Alfa

INTERVENTIONS:
Drug: Corifollitropin Alfa — late start (day 4) vs. corifollitropin-alfa standard start (day 2)

SUMMARY:
To compare the number of retrieved oocytes in the late start CF-alfa (day 4) versus standard CF-alfa protocols (day 2) in patients undergoing IVF. The primary analysis will be also performed in specific subgroups of patients: expected poor-responders, expected normal responders and expected hyper-responders

DETAILED DESCRIPTION:
The investigators hypothesize that:

1. CF-alfa late start (day 4) will show comparable efficacy in terms of number of retrieved oocytes versus standard CF-alfa (day 2) protocol. In certain groups of patients, CF-alfa late start might show differences in terms of efficacy such as in poor-responder patients.
2. CF-alfa late start (day 4) will obtain similar results in terms of vital pregnancy rates with a similar safety profile with respect to COS performed using CF-alfa standard administration (day 2) in expected normal, poor, or high responders.
3. Oocytes and embryos obtained using CF-alfa late start will have comparable morphological features and development potential than those obtained with CF-alfa standard.
4. The patients' satisfaction will possibly be higher using CF-alfa late start than with CF-alfa standard expecially in those patients who will not have the need to add further daily recFSH injections

ELIGIBILITY:
Inclusion Criteria:

* aged 18- 43 years
* Male or tubal infertility with indication for IVF treatment
* No PCOS
* No previous IVF treatments in the past two months
* No history of previous Ovarian Hyperstimulation Syndrome (OHSS)
* No previous IVF cycle with more than 30 growing follicles ≥ 11 mm
* Antral Follicle Count (AFC) <20
* No ovarian cyst nor malignant ovarian tumour, breast, uterus or central nervous cancer

Exclusion Criteria:

* AMH < 0.2 ng/ml
* Età > 43 anni

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
number of retrieved oocytes | 1 year
  To compare the number of retrieved oocytes in the late start CF-alfa (day 4) versus standard CF-alfa protocols (day 2) in patients undergoing IVF

CONTACTS AND LOCATIONS:
Locations (1):
- Physiopathology of Reproduction and IVF Unit, S. Anna Hospital, Torino, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Revelli A, Gennarelli G, Sestero M, Canosa S, Carosso A, Salvagno F, Pittatore G, Filippini C, Benedetto C. A prospective randomized trial comparing corifollitropin-alpha late-start (day 4) versus standard administration (day 2) in expected poor, normal, and high responders undergoing controlled ovarian stimulation for IVF. J Assist Reprod Genet. 2020 May;37(5):1163-1170. doi: 10.1007/s10815-020-01742-5. Epub 2020 Mar 18. PMID 32185595